CLINICAL TRIAL: NCT06513403
Title: Preliminary Study Using Artificial Intelligence Technology to Identify Differences in Facial Expressions Between Healthy People, Patients With Cognitive Decline, and Patients With Dementia
Brief Title: Preliminary Research Using Artificial Intelligence Technology to Identify Differences in Facial Expressions Between Healthy People, Patients With Cognitive Decline, and Patients With Dementia
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202405102RIN
Record Dates: First submitted 2024-07-17; First posted 2024-07-22 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-07

CONDITIONS: Artificial Intelligence Technology; Cognitive Decline; Dementia; Identify; Facial Expressions
Keywords: artificial intelligence technology; cognitive decline; dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Facial Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Through artificial intelligence technology, we have conducted a preliminary study aimed at identifying differences in facial expressions among healthy individuals, patients with cognitive decline, and dementia patients. This research offers a novel method and tool for dementia screening, contributing to effective strategies for dementia prevention in our country. By utilizing this approach, we can effectively delay the onset of disability, promote healthy aging among our elderly population, reduce the caregiving burden on individuals, families, and society, and lower medical expenses.

ELIGIBILITY:
Inclusion Criteria:

Age between 50 and 75 years.

* Experimental group:
* MCI group: CDR score of 0.5 or MMSE score between 20-25 (mild/early stage).
* Dementia group: CDR score greater than 1 or MMSE score between 10-19 (moderate/middle stage).
* Control group:
* Health group: MMSE score of 26 or above.
* Participants must be conscious and able to follow instructions.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Normal cognition group (Health): 20 participants
  * Mild cognitive impairment group (MCI): 20 participants
  * Dementia group: 20 participants
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Facial Expression Test | 2024/8/1-2025/10/31
  (A) Participants will sit in front of a computer screen and watch videos depicting positive (happy) or negative (sad) emotional stimuli. Each video will be less than 60 seconds long. (B) Participants will undergo the memory recall and calculation ability tests included in the MMSE. (C) While participants are undergoing the tests, video recording equipment will be used to observe and record the facial expression responses of the three groups.

CONTACTS AND LOCATIONS:
Locations (1):
- NTUH, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
The outcome of the current experiment is uncertain, so no decision has been made.